CLINICAL TRIAL: NCT02513966
Title: Decreased Consumption of Blood Components During Cardiac Surgery Procedures: Causes and Effects.
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s58228
Record Dates: First submitted 2015-07-13; First posted 2015-08-03 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2021-04

CONDITIONS: Blood Safety; Blood Transfusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is a decrease in the amount of blood components used during cardiac surgery in the last four years. As the hemovigilance team of the investigators' Hospital the investigators want to find out the causes and effects of this decrease.

ELIGIBILITY:
Inclusion Criteria:

* patient underwent cardiac surgery between 2010 and 2014 in UZ Leuven

Exclusion Criteria:

* patient without cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing cardiac surgery from 2010 untill 2014 in the University Hospitals of Leuven.
Sampling Method: Non-Probability Sample
Enrollment: 7835 (Actual)
Dates: Start 2015-07; Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
amount of blood use during Cardiac surgery | 5years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Devos, master, Study Chair — Universitaire Ziekenhuizen KU Leuven